CLINICAL TRIAL: NCT01041781
Title: A Randomized Phase III Double Blind Trial Evaluating Selective COX-2 Inhibition in COX-2 Expressing Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine Hydrochloride or Pemetrexed Disodium and Carboplatin With or Without Celecoxib in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommendation
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CALGB-30801; CALGB-30801; CDR0000662707 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Celecoxib; Gemcitabine; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride* IV on days 1 and 8 OR pemetrexed disodium* IV on day 1. Patients also receive carboplatin IV on day 1 and oral celecoxib twice daily on days 1-21.
  Interventions: Drug: carboplatin; Drug: celecoxib; Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium
- Arm II (Active Comparator): Patients receive gemcitabine hydrochloride* OR pemetrexed disodium* and carboplatin as in arm I. Patients also receive oral placebo twice daily on days 1-21.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium; Other: placebo

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: celecoxib — Given orally
  Arms: Arm I
Drug: gemcitabine hydrochloride — Given IV
Drug: pemetrexed disodium — Given IV
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium and celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving gemcitabine hydrochloride or pemetrexed disodium together with carboplatin is more effective with or without celecoxib in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying gemcitabine hydrochloride, pemetrexed disodium, and carboplatin to compare how well they work when given together with celecoxib or a placebo in treating patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To confirm the beneficial effect of gemcitabine hydrochloride or pemetrexed disodium in combination with carboplatin with or without celecoxib in patients with advanced non-small cell lung cancer that expresses COX-2.

Secondary

* To describe the response rate in patients treated with these regimens.
* To describe the distribution of progression-free survival (PFS) and overall survival of patients treated with these regimens.
* To compare the PFS of patients with COX-2 index ≥ 2 (adjusting for CYP2C9 genotype and celecoxib trough concentrations as covariates) treated with these regimens.
* To correlate urinary PGE-M level with COX-2 expression, COX-2 inhibition, and outcome.
* To evaluate the association between the -765G/C polymorphism in PTGS2 and COX-2 expression in non-small cell lung cancer specimens.
* To characterize a trough plasma celecoxib concentration which will be used as a measure of patient adherence to study treatment and which may be used in future studies for correlations with genotype and pharmacodynamic outcomes.

OUTLINE: This is a multicenter study. Patients are stratified according to gender, disease stage (IIIB vs IV), histology (squamous cell carcinoma vs non-squamous cell carcinoma), smoking status (never/former light smoker [defined as ≤ 10 pack years AND quit ≥ 1 year ago] vs smoker), and COX-2 expression status (COX-2 index ≥ 4 vs COX-2 index ≥ 2 but < 4). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride* IV on days 1 and 8 OR pemetrexed disodium* IV on day 1. Patients also receive carboplatin IV on day 1 and oral celecoxib twice daily on days 1-21.
* Arm II: Patients receive gemcitabine hydrochloride* OR pemetrexed disodium* and carboplatin as in arm I. Patients also receive oral placebo twice daily on days 1-21.
* NOTE: *Patients with squamous cell carcinoma receive gemcitabine hydrochloride; patients with non-squamous cell carcinoma receive pemetrexed disodium.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with responding or stable disease may continue to receive celecoxib or placebo alone in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood and urine sample collection periodically for correlative laboratory studies.

After completion of study therapy, patients are followed up every 2 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell carcinoma of the lung, including the following cell types:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Mixture of these types
* A tissue block must be available at the time of registration
* Tumor expresses COX-2 (COX-2 index ≥ 2)
* Stage IIIB disease with malignant pleural effusion, supraclavicular node involvement, or contralateral hilar node involvement OR stage IV disease

  * Patients with stage IIIB disease who are eligible for clinical trials that involve combined chemotherapy and chest irradiation are not eligible for this study
* Patients with stage IV disease are eligible
* Patients with recurrent disease, not amenable to (or refusing) a potentially "curative therapy," are eligible
* Measurable or non-measurable disease

  * Measurable disease is defined as lesions that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 2 cm with conventional techniques or as ≥ 1 cm with spiral CT scan
  * Non-measurable disease is defined as all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly nonmeasurable lesions, including any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients with symptomatic CNS metastases are eligible provided they received prior therapy (e.g., surgery, radiotherapy, or gamma knife), are neurologically stable, and are off steroids for ≥ 14 days before study entry

  * Patients with asymptomatic CNS metastases without associated edema, shift, or requirement for steroids or antiseizure medications may be eligible after discussion with the Study Chair
  * Patients should be off steroids at least 7 days before preregistration
* No leptomeningeal disease or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Granulocytes ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Creatinine clearance ≥ 45 mL/min
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.0 times upper limit of normal (ULN) (≤ 5.0 times ULN if liver metastases are present)
* Serum albumin ≥ 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* No "currently active" second malignancy other than non-melanoma skin cancer

  * Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at < 30% risk of relapse
* No known hypersensitivity to aspirin, NSAIDs, or sulfonamides
* No active ulcer disease

  * No history of gastrointestinal bleeding within the past three years
* None of the following cardiovascular conditions within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Serious uncontrolled cardiac arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
  * Symptomatic carotid artery or peripheral vascular disease
  * Deep vein thrombosis
  * Other significant thromboembolic event

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, immunotherapy, or other systemic therapy for non-small cell lung cancer, including adjuvant therapy
* At least 2 weeks since prior surgery and recovered
* At least 7 days since prior radiotherapy
* At least 14 days since prior NSAIDs (other than low-dose aspirin [≤ 325 mg daily]), including any of the following:

  * Celecoxib
  * Choline Mg
  * Trisalicylate (Trilisate®)
  * Ibuprofen (Advil® or Motrin®)
  * Naproxen (Aleve®, Naprosyn® or Anaprox®)
  * Etodolac (Lodine®)
  * Oxaprozin (Daypro®)
  * Diflunisal (Dolobid®)
  * Nabumetone (Relafen®)
  * Tolmetin (Tolectin®)
  * Valdecoxib (Bextra®)
* No chronic use of NSAIDs (i.e., > 4 weeks of daily use)

  * Patients on low-dose aspirin are eligible
* No other concurrent chemotherapy or hormonal therapy (other than megestrol acetate [Megace] for appetite stimulation)
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2010-02; Primary Completion 2017-01-17 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Edelman, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (399):
- United States (399):
  - Regional Medical Center, Anniston, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - NEA Medical Clinic - East Matthews, Jonesboro, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Feather River Hospital Cancer Center, Paradise, California
  - PCR Oncology, Pismo Beach, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - North Broward Medical Center, Deerfield Beach, Florida
  - Florida Hospital - Orlando, Orlando, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Helen G Nassif Community Cancer Center, Cedar Rapids, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - John R. Marsh Cancer Center at Washington County Hospital, Hagerstown, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers - Adrian, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Toledo Clinic Cancer Centers - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Veterans Administration/Harry S Truman Memorial Hospital, Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mercy-Springfield, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Administration New Jersey Health Care System, East Orange, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Toledo Clinic Cancers Centers - Maumee, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Centers of Southwest Oklahoma, LLC - Lawton, Lawton, Oklahoma
  - Mercy Clinic Oklahoma Communities Inc-Norman, Norman, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Mercy Clinic Oklahoma Communities Inc-Mercy Health Center, Oklahoma City, Oklahoma
  - Celilo Cancer Center at Mid-Columbia Medical Center, The Dalles, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System - Tacoma General Hospital, Tacoma, Washington
  - Saint Clare Hospital, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Minocqua Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Rice Lake Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Edelman MJ, Wang X, Hodgson L, Cheney RT, Baggstrom MQ, Thomas SP, Gajra A, Bertino E, Reckamp KL, Molina J, Schiller JH, Mitchell-Richards K, Friedman PN, Ritter J, Milne G, Hahn OM, Stinchcombe TE, Vokes EE; Alliance for Clinical Trials in Oncology. Phase III Randomized, Placebo-Controlled, Double-Blind Trial of Celecoxib in Addition to Standard Chemotherapy for Advanced Non-Small-Cell Lung Cancer With Cyclooxygenase-2 Overexpression: CALGB 30801 (Alliance). J Clin Oncol. 2017 Jul 1;35(19):2184-2192. doi: 10.1200/JCO.2016.71.3743. Epub 2017 May 10. PMID 28489511
- [Derived] Hamy AS, Tury S, Wang X, Gao J, Pierga JY, Giacchetti S, Brain E, Pistilli B, Marty M, Espie M, Benchimol G, Laas E, Lae M, Asselain B, Aouchiche B, Edelman M, Reyal F. Celecoxib With Neoadjuvant Chemotherapy for Breast Cancer Might Worsen Outcomes Differentially by COX-2 Expression and ER Status: Exploratory Analysis of the REMAGUS02 Trial. J Clin Oncol. 2019 Mar 10;37(8):624-635. doi: 10.1200/JCO.18.00636. Epub 2019 Jan 31. PMID 30702971

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Arm A: Celecoxib + Standard Chemotherapy): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1 and 8 (for those with squamous carcinoma) OR 500 mg/m^2 pemetrexed disodium IV on day 1 (for those with non-squamous carcinoma). Patients also receive (Squamous carcinoma patients: AUC=5.5 (Patient with prior chest radiotherapy should receive carboplatin at an AUC = 5.0); Non-squamous carcinoma patients: AUC=6.0) carboplatin IV on day 1 and 400 mg oral celecoxib twice daily on days 1-21. Patients may receive a maximum of 6 cycles of therapy (1 cycle = 21 days). Following 6 cycles of therapy, those patients with responding or stable disease will continue on the celecoxib/placebo until disease progression or unacceptable toxicity.
- Arm II (Arm B: Placebo + Standard Chemotherapy): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1 and 8 (for those with squamous carcinoma) OR 500 mg/m^2 pemetrexed disodium IV on day 1 (for those with non-squamous carcinoma). Patients also receive (Squamous carcinoma patients: AUC=5.5; Non-squamous carcinoma patients: AUC=6.0) carboplatin IV on day 1 and placebo twice daily on days 1-21. Patients may receive a maximum of 6 cycles of therapy (1 cycle = 21 days).
Period: Overall Study
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
Started | 154 | 158
Completed | 154 | 158
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy) | Total
Number analyzed (Participants) | 154 | 158 | 312
Age, Continuous [Median (Full Range); unit: years] | 64.0 [38.0 to 83.0] | 64.0 [36.0 to 89.0] | 64.0 [36.0 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 82 | 87 | 169
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 158 | 312

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time between randomization and disease relapse or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
Number analyzed (Participants) | 154 | 158
months | 5.16 [4.40 to 5.78] | 5.26 [4.40 to 6.08]
Statistical Analysis 1: Comparison: Arm I (Arm A: Celecoxib + Standard Chemotherapy) vs Arm II (Arm B: Placebo + Standard Chemotherapy); Test type: Superiority; p = 0.5346, Log Rank; Hazard Ratio (HR) = 1.076, 95% CI 2-sided [0.853 to 1.367]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time between randomization and death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Arm A: Celecoxib + Standard Chemotherapy): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1 and 8 (for those with squamous carcinoma) OR 500 mg/m^2 pemetrexed disodium IV on day 1 (for those with non-squamous carcinoma). Patients also receive (Squamous carcinoma patients: AUC=5.5; Non-squamous carcinoma patients: AUC=6.0) carboplatin IV on day 1 and 400 mg oral celecoxib twice daily on days 1-21.
- Arm II (Arm B: Placebo + Standard Chemotherapy): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1 and 8 (for those with squamous carcinoma) OR 500 mg/m^2 pemetrexed disodium IV on day 1 (for those with non-squamous carcinoma). Patients also receive (Squamous carcinoma patients: AUC=5.5; Non-squamous carcinoma patients: AUC=6.0) carboplatin IV on day 1 and placebo twice daily on days 1-21.
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
Number analyzed (Participants) | 154 | 158
months | 11.4 [9.46 to 14.06] | 12.5 [9.36 to 13.83]

3. Secondary Outcome: Response Rate
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients. Response rates (including complete and partial response) will be tested using Fisher's exact test
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
Number analyzed (Participants) | 154 | 158
percentage of patients | 40 [32 to 48] | 35 [27 to 43]

4. Secondary Outcome: Incidence of Toxicities as Assessed by NCI CTCAE v. 4.0
Description: The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment
Time Frame: Up to 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
Number analyzed (Participants) | 154 | 158
percentage of patients | 61.04 | 55.06

5. Secondary Outcome: Prognostic Value of Urinary Prostaglandin Metabolites (PGE-M) Levels for Worse PFS for Patients Who Had Baseline Urinary PGE-M Above/Below the First Quartile (Q1)
Description: Prognostic value of urinary prostaglandin metabolites (PGE-M) levels for worse PFS for patients who had baseline urinary PGE-M above/below the first quartile (Q1, 10.09). Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 5 years
Population: Patients on the placebo arm with urinary PGE-M evaluated at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- PGE-M < Q1: Patients with urinary PGE-M < Q1 (10.09) at baseline
- PGE-M >= Q1: Patients with urinary PGE-M >= Q1 (10.09) at baseline
Arm/Group | PGE-M < Q1 | PGE-M >= Q1
Number analyzed (Participants) | 27 | 78
months | 7.7 [4.40 to 13.14] | 4.9 [3.81 to 6.14]
Statistical Analysis 1: Comparison: PGE-M < Q1 vs PGE-M >= Q1; Test type: Superiority; p = 0.0049, Log Rank

6. Secondary Outcome: Prognostic Value of Urinary Prostaglandin Metabolites (PGE-M) Levels for Worse PFS for Patients Who Had Baseline Urinary PGE-M Above/Below the Median Quartile (Q2)
Description: prognostic value of urinary prostaglandin metabolites (PGE-M) levels for worse PFS for patients who had baseline urinary PGE-M above/below the median quartile (Q2, 15.38). Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 5 years
Population: Patients on the placebo arm with urinary PGE-M evaluated at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- PGE-M < Q2: Patients with urinary PGE-M < Q2 (15.38) at baseline
- PGE-M >= Q2: Patients with urinary PGE-M >= Q2 (15.38) at baseline
Arm/Group | PGE-M < Q2 | PGE-M >= Q2
Number analyzed (Participants) | 56 | 49
months | 6.2 [4.40 to 7.49] | 4.2 [3.42 to 5.78]
Statistical Analysis 1: Comparison: PGE-M < Q2 vs PGE-M >= Q2; Test type: Superiority; p = 0.0131, Log Rank

7. Secondary Outcome: Prognostic Value of Urinary Prostaglandin Metabolites (PGE-M) Levels for Worse PFS for Patients Who Had Baseline Urinary PGE-M Above/Below the Third Quartile (Q3)
Description: Prognostic value of urinary prostaglandin metabolites (PGE-M) levels for worse PFS for patients who had baseline urinary PGE-M above/below the median quartile (Q3, 27.86). Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 5 years
Population: Patients on the placebo arm with urinary PGE-M evaluated at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- PGE-M < Q3: Patients with urinary PGE-M < Q3 (27.86) at baseline
- PGE-M >= Q3: Patients with urinary PGE-M >= Q3 (27.86) at baseline
Arm/Group | PGE-M < Q3 | PGE-M >= Q3
Number analyzed (Participants) | 79 | 26
months | 6.0 [4.50 to 7.23] | 3.0 [1.77 to 5.09]
Statistical Analysis 1: Comparison: PGE-M < Q3 vs PGE-M >= Q3; Test type: Superiority; p = 0.0322, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events (AE) are collected each cycle during protocol therapy. AE forms are submitted until all protocol treatment related events have resolved or until non protocol treatment begins; Up to 5 years.
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed the study. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I (Arm A: Celecoxib + Standard Chemotherapy) | Arm II (Arm B: Placebo + Standard Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 15/146 | 9/148
Serious Adverse Events (participants affected / at risk) | 31/146 | 21/148
Other Adverse Events (participants affected / at risk) | 135/146 | 140/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Arm A: Celecoxib + Standard Chemotherapy) (N=146) | Arm II (Arm B: Placebo + Standard Chemotherapy) (N=148)
Anemia (Blood and lymphatic system disorders) | 22 (26) | 17 (19)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1)
Death NOS (General disorders) | 5 (5) | 4 (4)
Fatigue (General disorders) | 20 (23) | 15 (17)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 2 (2)
CPK increased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 8 (8) | 9 (10)
Platelet count decreased (Investigations) | 16 (17) | 12 (12)
White blood cell decreased (Investigations) | 2 (2) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)
Visceral arterial ischemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Arm A: Celecoxib + Standard Chemotherapy) (N=146) | Arm II (Arm B: Placebo + Standard Chemotherapy) (N=148)
Anemia (Blood and lymphatic system disorders) | 120 (566) | 123 (490)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 3 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (10) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 31 (47) | 23 (34)
Nausea (Gastrointestinal disorders) | 6 (7) | 11 (16)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 48 (79) | 32 (48)
Edema limbs (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 109 (423) | 115 (418)
Fever (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (12) | 4 (5)
Pain (General disorders) | 5 (5) | 4 (9)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 9 (12) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 2 (7)
Alkaline phosphatase increased (Investigations) | 2 (4) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (7)
Blood bilirubin increased (Investigations) | 5 (6) | 4 (6)
CD4 lymphocytes decreased (Investigations) | 2 (6) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (3) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 13 (17) | 16 (36)
Lymphocyte count increased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 66 (150) | 67 (138)
Platelet count decreased (Investigations) | 77 (207) | 78 (173)
Weight loss (Investigations) | 2 (3) | 2 (2)
White blood cell decreased (Investigations) | 15 (20) | 16 (26)
Anorexia (Metabolism and nutrition disorders) | 67 (160) | 64 (136)
Dehydration (Metabolism and nutrition disorders) | 8 (13) | 5 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (20) | 8 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 16 (37) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (10) | 4 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 12 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (7)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (10)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 (40) | 15 (20)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (6) | 8 (13)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes